CLINICAL TRIAL: NCT00135525
Title: Clinical Evaluation of BRL29060 A in Generalized Anxiety Disorder
Brief Title: Study Of Generalized Anxiety Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BRL29060A/856
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Anxiety Disorder; Anxiety Disorders
Keywords: Generalized Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paroxetine (Experimental): Fixed Dose (20 mg/day): The fixed dose of 20 mg/day was selected, because it is the recommended dose for the treatment of GAD in the US and other countries.
  Flexible Dose (20 - 40 mg/day): Overseas, the maximum dose in the treatment of GAD is 50 mg/day. However, 40 mg/day was selected as the maximum dose for this flexible dose session, because overseas clinical studies have indicated that paroxetine is sufficiently effective at doses of 20 - 40 mg/day and this is the dose range approved for depression/depressive episodes in Japan.
  Interventions: Drug: Paroxetine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paroxetine — Fixed Dose (20 mg/day): The fixed dose of 20 mg/day was selected, because it is the recommended dose for the treatment of GAD in the US and other countries.
  Flexible Dose (20 - 40 mg/day): Overseas, the maximum dose in the treatment of GAD is 50 mg/day. However, 40 mg/day was selected as the maximum dose for this flexible dose session, because overseas clinical studies have indicated that paroxetine is sufficiently effective at doses of 20 - 40 mg/day and this is the dose range approved for depression/depressive episodes in Japan.
  Arms: Paroxetine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy and safety in Generalized Anxiety Disorder patients

DETAILED DESCRIPTION:
This study was a multi-center, randomized, placebo-controlled, double-blinded (placebo run-in will be single-blinded), group comparison study.

Paroxetine 20mg/day (achieved via the starting dose of 10 mg/day for the first week) once daily, or placebo was orally administered once daily for 8 weeks (fixed dose was adopted in the Treatment phase) in patients with GAD.

For subjects who were classed as non-responders at Week 8, paroxetine at 30 to 40mg/day (once daily) or placebo (once daily) was orally administered with flexible titration regimen for 4 weeks (fixed dose was adopted in the Treatment phase). The subjects underwent a taper phase in case they received Paroxetine 40mg/day, paroxetine 30mg/day or placebo at treatment completion or study withdrawal. A follow-up examination was conducted after 1 to 5 weeks from the last dose of the investigational product.

The overall study duration requiring subject participation was 10 to 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Generalized Anxiety Disorder (GAD) according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria.
* Must give a written informed consent. But if the patient is under 20, both the patient himself/herself and his/her proxy consenter must give written informed consent.

Exclusion Criteria:

* Have the following conditions currently or diagnosed in the past 24 weeks:

Major Depressive Episode, Panic Disorder Without Agoraphobia, Panic Disorder With Agoraphobia, Social phobia/social anxiety disorder (SAD), Agoraphobia Without History of Panic Disorder, Posttraumatic Stress Disorder, Obsessive Compulsive Disorder, Anorexia Nervosa, Bulimia Nervosa, Dysthymic disorder

* Current or history of schizophrenia, bipolar disorder or cyclothymic disorder.
* Psychotherapy or cognitive behavioral therapy other than supportive psychotherapy.
* Current or history of substance abuse (alcohol or drugs) or substance in past 24 weeks.
* Taken St. John's Wort in past 4 weeks.
* Had electroconvulsive therapy (ECT) in past 12 weeks.
* Had psychotherapy or cognitive behavioral therapy other than supportive psychotherapy within 24 weeks.
* Women who are pregnant or lactating, who may be pregnant, or who plan for pregnancy by 30 days after the completion of final dose.
* Pose a suicidal threat or have attempted suicide in past 24 weeks.
* History of convulsive disorder (epilepsy, etc.).
* Significant unstable medical illness.
* Current or history of glaucoma.
* History or complication of cancer or malignant tumor.
* History of hypersensitivity to paroxetine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-05; Primary Completion 2005-10 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in the Hamilton Anxiety Scale (HAM-A) total score (at Week 8, last observation carried forward [LOCF]) | 8 Weeks

SECONDARY OUTCOMES:
Mean change from baseline in the HAM-A score (at Weeks 1, 2, 4 and 6); in the Severity of Illness (CGI SI) score; in the SDS and MADRS total scoreProportion of responders based on the Clinical Global Impression Global Improvement (CGI GI) score | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline